CLINICAL TRIAL: NCT05881629
Title: Early Diagnosis and Intervention for Fetal Malposition in Active Labor and Its Impact on Mode of Delivery: A Randomized Controlled Trial
Brief Title: Early Diagnosis and Intervention for Fetal Malposition in Active Labor and Its Impact on Mode of Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Kathryn Anderson, Resident physician, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015598-1
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Delivery Affecting Fetus; Labor Dystocia; Labor Complication
Keywords: fetal malposition; occiput posterior; occiput transverse
MeSH Terms: conditions — Dystocia; Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: Intervention group (side-lying position with peanut ball) versus control group (free position choice, no peanut ball)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Side-lying peanut ball group (Experimental): Participants randomized to this group will be asked to adopt a side-lying, lateral position on the ipsilateral side of the fetal spine. A peanut ball will be positioned between the participant's legs while in this position. They will be asked to maintain this position for 60 minutes.
  Interventions: Behavioral: Maternal position change to side-lying lateral with peanut ball
- Control group (Placebo Comparator): Participants randomized to this group will be able to adopt any position of their choosing during the 60-minute study period. They will not be able to use a peanut ball during this time.
  Interventions: Behavioral: Free maternal position

INTERVENTIONS:
Behavioral: Maternal position change to side-lying lateral with peanut ball — Participants will be assisted into a position lying on their side, specifically the same side as the fetal spine diagnosed by ultrasound. An inflated peanut ball will be positioned between the legs to open the pelvis. They will be asked to maintain the position for 60 minutes.
  Arms: Side-lying peanut ball group
Behavioral: Free maternal position — Participants will be asked to adopt any position of their choosing and to maintain it for 60 minutes. They will be asked to not use a peanut ball during the 60 minute study period.
  Arms: Control group

SUMMARY:
The goal of this randomized trial is to test if changing a person's position in labor can increase the chances of delivering their baby vaginally.

Specifically, it aims to answer the questions:

* In fetuses who are facing upwards (occiput posterior, OP) or sideways (occiput transverse, OT) during labor, does changing the patient's position during active labor to a side-lying posture with a peanut ball increase the chances of them having a successful, spontaneous vaginal delivery?
* Does changing the patient's position in active labor affect the position of the baby at the time of delivery?
* Do intentional position changes in labor impact patient-perceived autonomy during their labor and delivery experience?

Participants will:

* Receive an ultrasound during labor to determine the position of their baby
* Be asked to adopt a specific position in labor (side-lying with peanut ball) if they are randomized to the study group
* Receive additional ultrasounds during labor to assess their baby's position
* Fill out a questionnaire about their labor experience following the delivery of their baby

DETAILED DESCRIPTION:
In this randomized trial, the investigators aim to evaluate the effects of early ultrasound diagnosis and active management of fetal malposition during the first stage of labor. Specifically, the investigators will compare the modified Sims (side-lying) position ipsilateral to fetal spine with the addition of a peanut ball versus free maternal position choice in occiput posterior (OP) or occiput transverse (OT) fetuses diagnosed by ultrasound during active labor, defined as greater than 6cm cervical dilation. The primary outcome will be operative delivery rates, defined as either cesarean delivery or instrumental vaginal delivery with vacuum or forceps. The investigators will also assess rates of spontaneous rotation to occiput anterior (OA) position at complete dilation and at delivery, as well as the impact of the position changes on the patient's labor experience and their perceived autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age >18
* Term gestation (>37 weeks)
* Singleton pregnancy
* Spontaneous or induced active labor (cervical dilation 6-9cm)
* Epidural anesthesia
* Cephalic fetal presentation, OP/OT position diagnosed by bedside ultrasound
* Continuous external fetal monitoring
* Ability to consent

Exclusion Criteria:

* Multiple gestations
* Unanesthetized labor
* Known fetal anomalies
* Known intrauterine fetal demise
* Inability to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Operative Delivery Rate | Enrollment in active labor through delivery, on average 12 hours
  The combined rate of cesarean and instrumental vaginal deliveries in each study group

SECONDARY OUTCOMES:
Rotation at Complete Dilation | Enrollment in active labor through delivery, on average 12 hours
  The percent of fetuses that rotate to facing downwards (occiput anterior) at the time of complete cervical dilation (10cm) in each study group
Rotation at Delivery | Enrollment in active labor through delivery, on average 12 hours
  The percent of fetuses that rotate to facing downwards (occiput anterior, OA) at the time of delivery in each study group
Duration of Active Second Stage | Onset of second stage of labor to delivery, up to 4 hours
  The mean amount of time spent pushing during the second stage of labor in each group (measured in minutes)
Estimated Blood Loss | Time of delivery to 24 hours postpartum
  The mean amount of blood loss incurred at delivery in each study group (measured in mL)
Degree of Laceration following Delivery | Time of delivery to admission to postpartum unit, on average 2 hours
  The percent of each degree of vaginal laceration (first, second, third, fourth) sustained during vaginal delivery in each study group
Score on Labor Agentry Scale | Time of delivery to discharge from hospital, on average 2 days
  The mean score on the validated Labor Agentry Scale (LAS) in each study group, which measures the degree that the participant felt in control during their labor process. Possible total scores for the Labor Agentry Scale range from 10 (rarely felt in control) to 70 (almost always felt in control).
Apgar Scores | Time of delivery to 5 minutes postpartum
  Mean Apgar Score at 1 and 5 minutes for fetuses delivered in each study group
Neonatal Intensive Care Unit (NICU) Admission | Time of delivery to up to 6 weeks postpartum
  Rates of NICU admission following delivery in each study group

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Gimovsky, MD, Principal Investigator — Women and Infant's Hospital of Rhode Island
Locations (1):
- Women and Infant's Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No